CLINICAL TRIAL: NCT02806193
Title: Global Cardiovascular Magnetic Resonance Registry
Brief Title: Global CMR Registry
Acronym: GCMR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Society for Cardiovascular Magnetic Resonance (Other)
Responsible Party: Sponsor
Other Study IDs: SCMR_GRANT_001
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular; cardiac; MRI; CMR; CT; ECG; magnetic resonance; imaging
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiovascular Magnetic Resonance Imaging: Cardiovascular imaging techniques (other subsidiary techniques such as CT and ECG will also be followed)
  Interventions: Procedure: Cardiovascular Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Cardiovascular Magnetic Resonance Imaging — Cardiac magnetic resonance imaging (CMR) has emerged as both a remarkably powerful diagnostic and prognostic tool for the assessment of cardiovascular disease. The high spatial resolution of CMR and the ability to characterize soft tissue provides the opportunity for unique diagnostic assessment of a myriad of cardiac pathology, including ischemic heart disease (IHD), preoperative assessment, intra- cardiac mass and thrombus, pericardial disease, valvular heart disease, and cardiomyopathy evaluation.
  Between individual CMR programs, GCMR will offer information useful in assessing the differences in protocol, performance, and clinical adaptation by varying geographic regions, institutional environments, and expertise. Such an assessment is critical for uncovering possible reasons for disparities in performance and obtaining opportunities for advancement.

SUMMARY:
The Global CMR Registry aims to promote collaboration of CMR sites worldwide in setting imaging and reporting standards, assessing its diagnostic impact on patient care, and determining the cost-effectiveness of CMR imaging. It will be the largest collective body of evidence reflecting the current clinical applications in patient care, which healthcare payers and governing bodies alike can depend on when metrics such as testing appropriateness, common indications, and diagnostic effectiveness are called for. It will also be able to reflect any changes in patient impact from CMR over time as technical development evolves. Furthermore, it will allow an assessment of improvements in diagnostic and therapeutic thinking, risk stratification, and cost-effectiveness relevant to current patient management.

DETAILED DESCRIPTION:
A global CMR registry can be a crucial infrastructure of our CMR community that has many benefits. First, it is the largest collective body of evidence reflecting the current clinical applications in patient care, which healthcare payers and governing bodies alike can depend on when metrics such as testing appropriateness, common indications, and diagnostic effectiveness are needed. Second, it reflects any change in patient impact from CMR over time as technical developments evolve. Third, it allows an assessment for improvement of diagnostic and therapeutic evaluation, risk stratification, and cost-effectiveness analysis relevant to patient management.

Some practical questions that a global CMR registry may be able ot address include:

1. Variations in CMR protocols within specific clinical indications
2. Variations in CMR post-processing, analysis, and reporting
3. Practice adherence to appropriateness criteria and guidelines
4. Clinical effectiveness of CMR over a long period of clinical application and/or technological advance
5. Differences in CMR utility across centers, regions, or countries

The data collection process will be a collective effort on part of specialized health professionals across various CMR sites worldwide. All of the data will be extracted from existing registries and databases. Health professionals in the U.S. and abroad will first upload patient data and images onto the registry/database that they currently use. Then if they choose to, they can transmit relevant patient de-identified data onto the global registry using a user-friendly web interface. CMR sites without a database will be invited to use CMR Cooperative or REDCAP. De-identified data (usually submitted in excel or CSV format) will be harmonized and uploaded to the registry website (www.gcmr-scmr.org), which is a firewall and password-protected database that resides at an IT vendor (Center for Systems Biology at Massachusetts General Hospital) in Boston, Massachusetts. The pooled data will be used for retrospective analysis/research approved by the GCMR steering committee and SCMR.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular disease, underwent CMR, CT, or ECG

Exclusion Criteria:

* Patients who are 90 years and older

Max Age: 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry data will be collected from patients of various clinical CMR sites that have agreed to contribute their data to the registry.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | Mortality will be tracked through study completion, for each year
  death from various causes including cardiovascular death
Heart Failure | Through study completion, for each year
  heart failure development or worsening of heart failure
Acute myocardial infarction | Through study completion, for each year

SECONDARY OUTCOMES:
Cardiac Intervention (Implantable cardioverter-defibrillator or ICD) | Through study completion, for each year
Cardiac Intervention (pacemakers) | Through study completion, for each year
Cardiac Intervention (cardiac surgery) | Through study completion, for each year
Cardiac Intervention (coronary revascularization) | Through study completion, for each year

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Y. Kwong, MD, MPH, Study Chair — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Participating sites will send relevant de-identified to the data management team for harmonization. The aggregate data will be used for retrospective analyses and research. Researchers requesting data access for either grant proposals or sub-studies will be required to submit a proposal to the GCMR steering committee (composed of various experts in the CMR community) for approval.
  If approved, data access will be given to the researchers for a specific time period determined by the magnitude of the work involved, and only for the purposes of the grant proposal or sub-study.

REFERENCES:
- [Derived] Global Cardiovascular Magnetic Resonance Registry (GCMR) Investigators; Kwong RY, Petersen SE, Schulz-Menger J, Arai AE, Bingham SE, Chen Y, Choi YL, Cury RC, Ferreira VM, Flamm SD, Steel K, Bandettini WP, Martin ET, Nallamshetty L, Neubauer S, Raman SV, Schelbert EB, Valeti US, Cao JJ, Reichek N, Young AA, Fexon L, Pivovarov M, Ferrari VA, Simonetti OP. The global cardiovascular magnetic resonance registry (GCMR) of the society for cardiovascular magnetic resonance (SCMR): its goals, rationale, data infrastructure, and current developments. J Cardiovasc Magn Reson. 2017 Jan 20;19(1):23. doi: 10.1186/s12968-016-0321-7. PMID 28187739